CLINICAL TRIAL: NCT02906579
Title: An Open-label, Phase 2a Trial to Evaluate the Effect of Escalating Doses of IW-1973 on Tolerability, Endothelial Function, and Hemodynamics in Patients With Stable Type 2 Diabetes and Hypertension
Brief Title: A Phase 2 Trial of IW-1973, A Stimulator of Soluble Guanylate Cyclase (sGC), in Patients With Stable Type 2 Diabetes and Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1973-201
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — praliciguat

ARMS (1):
- IW-1973 (Experimental): Placebo taken once daily Day 1-Day 3; 10 mg IW-1973 take once daily Day 4-Day 6; 20 mg IW-1973 taken once daily Day 7-Day 9; 30 mg IW-1973 taken once daily Day 10-Day 12; 40 mg IW-1973 taken once daily Day 13-Day 15; 50 mg IW-1973 taken once daily Day 16-Day 18
  Interventions: Drug: Matching Placebo; Drug: IW-1973

INTERVENTIONS:
Drug: Matching Placebo
Drug: IW-1973

SUMMARY:
To evaluate the impact of escalating doses of IW-1973 on endothelial function [using EndoPAT to measure fingertip small vessel pulse volume], blood pressure (BP), and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ambulatory male or female
* Patient's body mass index score is >20 and <40 kg/m2 at the Screening Visit
* Women of childbearing potential must have a negative pregnancy test at the time of check-in and must agree to use double-barrier contraception throughout the duration of the study
* Patient's health is stable with no clinically significant findings on a physical examination
* Patient has type 2 (ie adult onset) diabetes mellitus diagnosed by a physician or nurse practitioner > 6 months before the Screening Visit, and an entry HbA1c that does not mandate prompt intervention for improved control
* Patient has hypertension diagnosed by a physician or nurse practitioner > 6 months before the Screening Visit and BP within the protocol's acceptable range
* Patients must be on a stable regimen for glycemic control, and a stable regimen for hypertension control that includes an angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB)
* Patient has abnormal endothelial function measured by the EndoPAT
* Other inclusion criteria per protocol

Exclusion Criteria:

* Patient has a clinically significant active or unstable medical condition that, in the opinion of the Investigator, would preclude trial participation
* Patient is on medication(s) that when co-administered with a soluble guanylate cyclase (sGC) stimulator, could increase the risk of hypotension
* Patient has evidence of severe or active end-organ damage attributable to diabetes
* Patient has severe renal insufficiency, has undergone renal transplantation, or has planned renal transplantation
* Other exclusion criteria per protocol

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Unit, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Once-daily study drug for 18 days: placebo for 3 days and escalating doses of IW-1973 for 15 days (10 mg, 20 mg, 30 mg, 40 mg, 50 mg for 3 days each).
Period: Overall Study
Arm/Group | All Participants
Started | 11
Completed Cycle 1 (Placebo) | 11
Completed Cycle 2 (10 mg IW-1973) | 11
Completed Cycle 3 (20 mg IW-1973) | 11
Completed Cycle 4 (30 mg IW-1973) | 10
Completed Cycle 5 (40 mg IW-1973) | 9
Completed Cycle 6 (50 mg IW-1973) | 9
Completed | 9
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6
  Black or African American | 5
Study Baseline: Supine systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Study baseline is defined as the Day -1 assessment.
  mmHg | 136.3 (12.9)
Study Baseline: Supine diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Study baseline is defined as the Day -1 assessment.
  mmHg | 80.4 (5.9)
Study Baseline: Pulse [Mean (Standard Deviation); unit: beats per minute] — Study baseline is defined as the Day -1 assessment.
  beats per minute | 72.0 (15.9)
Study Baseline: Cholesterol, Glucose, HDL-C, LDL-C, Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Study baseline is defined as the Day -1 assessment.
  mg/dL
    Cholesterol | 185.0 (44.9)
    Glucose | 143.27 (34.34)
    High-density lipoprotein cholesterol (HDL-C) | 50.27 (14.11)
    Low-density lipoprotein cholesterol (LDL-C) | 107.45 (36.74)
    Triglycerides | 137.73 (54.23)
Study Baseline: Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase [Mean (Standard Deviation); unit: U/L] — Study baseline is defined as the Day -1 assessment.
  U/L
    GGT | 36.2 (28.4)
    Lactate Dehydrogenase | 163.1 (30.7)
Study Baseline: Hemoglobin A1c [Mean (Standard Deviation); unit: percent] — Study baseline is defined as the Day -1 assessment.
  percent | 7.67 (1.33)
Study Baseline: Insulin [Mean (Standard Deviation); unit: μIU/mL] — Study baseline is defined as the Day -1 assessment.
  μIU/mL | 17.50 (12.17)
Study Baseline: Respiratory Rate [Mean (Standard Deviation); unit: breaths/min] — Study baseline is defined as the Day -1 assessment.
  breaths/min | 16.4 (2.2)
Study Baseline: Temperature [Mean (Standard Deviation); unit: degrees celcius] — Study baseline is defined as the Day -1 assessment.
  degrees celcius | 36.68 (0.21)
Study Baseline: Weight [Mean (Standard Deviation); unit: kg] — Study baseline is defined as the Day -1 assessment.
  kg | 91.08 (11.58)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Deaths, and Discontinuations Due to TEAEs
Description: An adverse event (AE) is any untoward medical occurrence, which does not necessarily have to have a causal relationship with study treatment. An SAE is defined as any AE occurring at any dose that results in any of the following outcomes: death; life-threatening; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical events. TEAEs are defined as those AEs that started or worsened in severity after the initiation of study drug administration.
Time Frame: From first dose of study drug through end of trial (Day 46 [±3 days])
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Count of Participants; unit: Participants
Groups:
- Control: Placebo taken once daily Day 1-Day 3
- 10 mg IW-1973: 10 mg IW-1973 take once daily Day 4-Day 6
- 20 mg IW-1973: 20 mg IW-1973 taken once daily Day 7-Day 9
- 30 mg IW-1973: 30 mg IW-1973 taken once daily Day 10-Day 12
- 40 mg IW-1973: 40 mg IW-1973 taken once daily Day 13-Day 15
- 50 mg IW-1973: 50 mg IW-1973 taken once daily Day 16-Day 18
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
Participants
  ≥1 TEAE | 3 | 3 | 2 | 4 | 3 | 2
  SAE | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0
  Discontinuations (DCs) due to AEs | 0 | 0 | 1 | 0 | 0 | 0
  DCs Due to Trough Blood Pressure Decline | 0 | 0 | 1 | 1 | 0 | 0

2. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Cholesterol, Glucose, HDL-C, LDL-C, and Triglycerides at Discharge Day (Day 19)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 11
mg/dL
  Cholesterol: Day 19/Discharge | 141.7 (39.6)
  Cholesterol: Change at Day 19/Discharge | -43.3 (35.1)
  Glucose: Day 19/Discharge | 116.82 (25.43)
  Glucose: Change at Day 19/Discharge | -26.45 (25.25)
  HDL-C: Day 19/Discharge | 44.36 (10.74)
  HDL-C: Change at Day 19/Discharge | -5.91 (7.73)
  LDL-C: Day 19/Discharge | 73.09 (34.69)
  LDL-C: Change at Day 19/Discharge | -34.36 (28.88)
  Triglycerides: Day 19/Discharge | 121.73 (46.10)
  Triglycerides: Change at Day 19/Discharge | -16.00 (42.45)

3. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Cholesterol, Glucose, HDL-C, LDL-C, and Triglycerides at Follow-Up (Day 32)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 11
mg/dL
  Cholesterol: Day 32/Follow-Up | 183.1 (48.6)
  Cholesterol: Change at Day 32/Follow-Up | -1.9 (27.1)
  Glucose: Day 32/Follow-Up | 154.27 (48.54)
  Glucose: Change at Day 32/Follow-Up | 11.00 (41.47)
  HDL-C: Day 32/Follow-Up | 48.18 (10.32)
  HDL-C: Change at Day 32/Follow-Up | -2.09 (6.88)
  LDL-C: Day 32/Follow-Up | 107.27 (42.11)
  LDL-C: Change at Day 32/Follow-Up | -0.18 (23.84)
  Triglycerides: Day 32/Follow-Up | 138.09 (46.26)
  Triglycerides: Change at Day 32/Follow-Up | 0.36 (52.94)

4. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase at Discharge Day (Day 19)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | All Participants
Number analyzed (Participants) | 11
U/L
  GGT: Day 19/Discharge | 28.3 (17.2)
  GGT: Change at Day 19/Discharge | -7.9 (15.9)
  Lactate Dehydrogenase: Day 19/Discharge | 135.7 (18.2)
  Lactate Dehydrogenase: Change at Day 19/Discharge | -27.4 (21.2)

5. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in GGT and Lactate Dehydrogenase at Follow-Up (Day 32)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | All Participants
Number analyzed (Participants) | 11
U/L
  GGT: Day 32/Follow-Up | 53.6 (83.9)
  GGT: Change at Day 32/Follow-Up | 17.5 (67.8)
  Lactate Dehydrogenase: Day 32/Follow-Up | 171.6 (55.2)
  Lactate Dehydrogenase: Change at Day 32/Follow-Up | 8.5 (46.4)

6. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Hemoglobin A1c at Discharge Day (Day 19)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Participants
Number analyzed (Participants) | 11
percent
  Discharge Day (Day 19) | 7.27 (1.53)
  Change at Discharge Day (Day 19) | -0.40 (0.54)

7. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Hemoglobin A1c at Follow-Up (Day 32)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | All Participants
Number analyzed (Participants) | 11
percent
  Follow-Up (Day 32) | 7.54 (1.49)
  Change at Follow-Up (Day 32) | -0.14 (0.49)

8. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Insulin at Discharge Day (Day 19)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | All Participants
Number analyzed (Participants) | 11
µIU/mL
  Discharge Day (Day 19) | 17.45 (14.20)
  Change at Discharge Day (Day 19) | -0.05 (5.31)

9. Primary Outcome: Certain Clinical Chemistry Laboratory Parameters: Overall Changes From Study Baseline in Insulin at Follow-Up (Day 32)
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Baseline, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | All Participants
Number analyzed (Participants) | 11
µIU/mL
  Follow-Up (Day 32) | 23.81 (18.81)
  Change at Follow-Up (Day 32) | 6.31 (11.18)

10. Primary Outcome: Change From Time-Matched Baseline in Fasting Blood Glucose on Day 2 of Each Dose Cycle
Description: Time-matched baseline is defined as the corresponding assessment on Day 2 of the placebo cycle.
  Baseline is designated per protocol as Day 2 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment). To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 2 of each IW-1973 dose are presented as the second row of data.
Time Frame: Time-Matched Baseline (Day 2 Placebo Cycle), Day 2 of Each Dose Cycle (Days 5, 8, 11, 14, 17)
Population: Pharmacodynamic (PD) Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
mg/dL
  Time-Matched Baseline | 142.3 (32.6) | 142.3 (32.6) | 144.1 (33.8) | 147.7 (33.8) | 147.7 (33.8)
  Cycle Day 2 Change | -12.0 (10.3) | -13.4 (9.9) | -21.1 (16.0) | -24.3 (16.9) | -25.3 (15.9)

11. Primary Outcome: Change From Time-Matched Baseline in Serum Insulin on Day 2 of Each Dose Cycle
Description: as for outcome 10
Time Frame: Time-Matched Baseline (Day 2 Placebo Cycle), Day 2 of Each Dose Cycle (Days 5, 8, 11, 14, 17)
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
µIU/mL
  Time-Matched Baseline | 17.35 (10.70) | 17.35 (10.70) | 17.37 (11.28) | 14.32 (6.21) | 14.32 (6.21)
  Cycle Day 2 Change | 0.20 (5.04) | -0.40 (6.26) | -2.61 (3.11) | -2.49 (5.65) | -2.70 (4.20)

12. Primary Outcome: Number of Participants With Notable Changes in Post Baseline Vital Signs Values
Description: Supine systolic blood pressure (SSBP):
  ≥ 180 mmHg and increase (↑) from baseline (BL) ≥ 30 mmHg; ≤ 90 mmHg and decrease (↓) from BL ≥ 30 mmHg.
  Supine Diastolic Blood Pressure (SDBP):
  ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg; ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg.
  Supine pulse rate (SPR):
  ≥ 110 beats per minute (bpm) and ↑ from BL ≥ 20 bpm; ≤ 50 bpm and ↓ from BL ≥ 20 bpm.
  Standing systolic blood pressure (StSBP):
  ≥ 180 mmHg and increase (↑) from baseline (BL) ≥ 30 mmHg; ≤ 90 mmHg and decrease (↓) from BL ≥ 30 mmHg.
  Standing Diastolic Blood Pressure (StDBP):
  ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg; ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg.
  Standing pulse rate (StPR):
  ≥ 110 beats per minute (bpm) and ↑ from BL ≥ 20 bpm; ≤ 50 bpm and ↓ from BL ≥ 20 bpm.
Time Frame: Up to Day 32
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
Participants
  SSBP: ≥ 180 mmHg and ↑ from BL ≥ 30 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  SSBP: ≤ 90 mmHg and ↓ from BL ≥ 30 mmHg | 0 | 0 | 1 | 2 | 0 | 0
  SDBP: ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  SDBP: ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  SPR: ≥ 110 bpm and ↑ from BL | 0 | 0 | 0 | 0 | 0 | 0
  SPR: ≤ 50 bpm and ↓ from BL ≥ 20 bpm | 0 | 0 | 0 | 0 | 0 | 0
  StSBP: ≥ 180 mmHg and ↑ from BL ≥ 30 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  StSBP: ≤ 90 mmHg and ↓ from BL ≥ 30 mmHg | 0 | 0 | 0 | 0 | 1 | 0
  StDBP: ≥ 105 mmHg and ↑ from BL ≥ 20 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  StDBP: ≤ 50 mmHg and ↓ from BL ≥ 20 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  StPR: ≥ 120 bpm and ↑ from BL | 0 | 0 | 0 | 0 | 0 | 0
  StPR: ≤ 50 bpm and ↓ from BL ≥ 20 bpm | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Notable Post Baseline Orthostatic Vital Signs Values
Description: Systolic blood pressure (SBP): Decrease of > 20 mmHg from supine to standing Diastolic blood pressure (DBP): Decrease of > 10 mmHg from supine to standing Pulse rate (PR): Increase of > 20 bpm from supine to standing.
Time Frame: Up to Day 32
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
Participants
  SBP: Decrease of > 20 mmHg, supine to standing | 0 | 0 | 0 | 0 | 0 | 0
  DBP: Decrease of > 10 mmHg from supine to standin | 0 | 0 | 1 | 0 | 1 | 0
  PR: Increase of > 20 bpm from supine to standing | 3 | 4 | 3 | 5 | 3 | 3

14. Primary Outcome: Change From Baseline Over Time in Respiratory Rate
Time Frame: Baseline, Day 19, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | All Participants
Number analyzed (Participants) | 11
breaths/min
  Change at Day 19/Discharge | -0.7 (1.8)
  Change at Day 32/Follow-Up | -1.5 (2.7)

15. Primary Outcome: Change From Baseline Over Time in Temperature
Time Frame: Baseline, Day 19, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: degrees celcius
Arm/Group | All Participants
Number analyzed (Participants) | 11
degrees celcius
  Change at Day 19/Discharge | 0.12 (0.19)
  Change at Day 32/Follow-Up | -0.03 (0.20)

16. Primary Outcome: Change From Baseline Over Time in Weight
Time Frame: Baseline, Day 19, Day 32
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | All Participants
Number analyzed (Participants) | 11
kg
  Change at Day 19/Discharge | -3.47 (2.16)
  Change at Day 32/Follow-Up | -1.40 (1.61)

17. Primary Outcome: Number of Participants With Clinically Significant Findings or Shifts in Baseline in Electrocardiograms (ECGs)
Time Frame: Study Baseline, Cycle Day 1: 0 (≤ 15m) predose; 1h, 4h (± 15m) postdose; Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 11
Participants | 0

18. Primary Outcome: Number of Participants With Clinically Significant Findings or Shifts in Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF)
Time Frame: Study Baseline, Cycle Day 1: 0 (≤ 15m) predose; 1h, 4h (± 15m) postdose; Day 19
Population: Safety Population: all participants who received ≥1 dose of study drug, grouped according to actual study drug taken.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Change From Study Baseline Over Time in Supine Pulse
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: Study Baseline; Cycle Day 1, 0 h; Cycle Day 1, 1 h; Cycle Day 1, 2 h; Cycle Day 1, 4 h; Cycle Day 1, 8 h; Cycle Day 1, 12 h; Cycle Day 3, 0 h; Cycle Day 3, 1 h; Cycle Day 3, 2 h; Cycle Day 3, 8 h
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
bpm
  Study Baseline | 72.0 (15.9) | 72.0 (15.9) | 72.0 (15.9) | 72.7 (16.6) | 73.2 (17.5) | 73.2 (17.5)
  Change at Cycle Day 1, 0 h | -5.5 (7.6) | -6.5 (11.6) | -5.8 (11.1) | -7.2 (11.0) | -4.9 (12.1) | -6.3 (13.7)
  Change at Cycle Day 1, 1 h | -0.1 (8.7) | -1.9 (9.8) | 1.7 (12.7) | 5.7 (12.7) | 1.0 (9.4) | 4.8 (12.1)
  Change at Cycle Day 1, 2 h | -1.8 (7.6) | 3.4 (8.9) | 6.3 (11.7) | 11.9 (14.1) | 13.9 (10.9) | 9.0 (12.1)
  Change at Cycle Day 1, 4 h | -3.5 (9.4) | -2.2 (10.7) | 1.7 (9.5) | 0.7 (10.6) | 3.7 (7.5) | 0.2 (8.8)
  Change at Cycle Day 1, 8 h | -3.2 (9.7) | 2.1 (12.3) | 0.8 (10.2) | -1.4 (9.3) | -1.7 (11.7) | -0.2 (8.9)
  Change at Cycle Day 1, 12 h | -2.3 (8.4) | 4.1 (10.4) | 2.9 (9.6) | 0 (9.4) | 3.2 (12.9) | 0.8 (10.2)
  Change at Cycle Day 3, 0 h | -4.1 (11.7) | -6.2 (10.7) | -5.1 (11.2) | -5.4 (10.8) | -6.8 (12.2) | -6.3 (11.4)
  Change at Cycle Day 3, 1 h | -1.8 (9.3) | 3.9 (11.9) | 5.5 (11.7) | 6.1 (8.4) | 8.8 (15.2) | 10.0 (13.2)
  Change at Cycle Day 3, 2 h | 2.0 (9.1) | 4.5 (11.3) | 7.2 (8.9) | 9.1 (10.7) | 11.1 (12.6) | 11.6 (13.1)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | -1.0 (11.2) | 0.6 (9.3) | -1.6 (11.7) | -1.2 (7.8) | -0.3 (11.4) | 4.2 (14.8)

20. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in Supine Pulse
Description: Time-matched baseline for each timepoint is defined as the corresponding assessment during the placebo cycle.
  Baseline is designated per protocol as Day 1 or 3 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 1 or 3 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 1, 0 h; Cycle Day 1, 1 h; Cycle Day 1, 2 h; Cycle Day 1, 4 h; Cycle Day 1, 8 h; Cycle Day 1, 12 h; Cycle Day 3, 0 h; Cycle Day 3, 1 h; Cycle Day 3, 2 h; Cycle Day 3, 8 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
bpm
  Time Matched Baseline (Cycle Day 1, 0 h) | 66.5 (10.8) | 66.5 (10.8) | 66.7 (11.3) | 67.0 (12.0) | 67.0 (12.0)
  Change at Cycle Day 1, 0 h | -1.1 (5.5) | -0.4 (5.2) | -1.2 (5.7) | 1.3 (7.0) | -0.1 (8.4)
  Time Matched Baseline (Cycle Day 1, 1 h) | 71.9 (12.6) | 71.9 (12.6) | 72.6 (13.0) | 73.4 (13.5) | 73.4 (13.5)
  Change at Cycle Day 1, 1 h | -1.8 (3.2) | 1.8 (5.0) | 5.8 (4.7) | 0.8 (4.5) | 4.6 (4.3)
  Time Matched Baseline (Cycle Day 1, 2 h) | 70.2 (11.7) | 70.2 (11.7) | 70.8 (12.2) | 71.8 (12.5) | 71.8 (12.5)
  Change at Cycle Day 1, 2 h | 5.2 (4.3) | 8.1 (6.7) | 13.8 (7.2) | 15.3 (7.2) | 10.4 (5.8)
  Time Matched Baseline (Cycle Day 1, 4 h) | 68.5 (10.4) | 68.5 (10.4) | 68.3 (10.9) | 68.4 (11.6) | 68.4 (11.6)
  Change at Cycle Day 1, 4 h | 1.3 (6.2) | 5.2 (7.7) | 5.1 (7.5) | 8.4 (6.8) | 5.0 (4.5)
  Time Matched Baseline (Cycle Day 1, 8 h) | 68.8 (10.9) | 68.8 (10.9) | 68.6 (11.5) | 68.9 (12.1) | 68.9 (12.1)
  Change at Cycle Day 1, 8 h | 5.3 (6.3) | 4.0 (3.8) | 2.7 (4.8) | 2.7 (5.8) | 4.1 (4.9)
  Time Matched Baseline (Cycle Day 1, 12 h) | 69.7 (11.5) | 69.7 (11.5) | 70.0 (12.1) | 70.2 (12.8) | 70.2 (12.8)
  Change at Cycle Day 1, 12 h | 6.4 (6.3) | 5.2 (5.9) | 2.7 (4.0) | 6.2 (7.3) | 3.8 (5.2)
  Time Matched Baseline (Cycle Day 3, 0 h) | 67.9 (11.9) | 67.9 (11.9) | 66.6 (11.7) | 67.1 (12.3) | 67.1 (12.3)
  Change at Cycle Day 3, 0 h | -2.1 (4.2) | -1.0 (6.4) | 0.7 (6.1) | -0.7 (2.9) | -0.2 (3.8)
  Time Matched Baseline (Cycle Day 3, 1 h) | 70.2 (13.6) | 70.2 (13.6) | 70.6 (14.3) | 71.2 (15.0) | 71.2 (15.0)
  Change at Cycle Day 3, 1 h | 5.7 (8.6) | 7.4 (9.9) | 8.2 (5.4) | 10.8 (6.9) | 12.0 (6.4)
  Time Matched Baseline (Cycle Day 3, 2 h): number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Time Matched Baseline (Cycle Day 3, 2 h) | 73.8 (15.0) | 73.8 (15.0) | 74.2 (15.9) | 75.6 (16.4) | 75.6 (16.4)
  Change at Cycle Day 3, 2 h: number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Change at Cycle Day 3, 2 h | 3.7 (6.2) | 5.1 (6.2) | 8.0 (6.3) | 10.3 (6.9) | 10.4 (8.3)
  Time Matched Baseline (Cycle Day 3, 8 h): number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Time Matched Baseline (Cycle Day 3, 8 h) | 71.0 (12.9) | 71.0 (12.9) | 69.8 (14.1) | 70.8 (14.1) | 70.8 (14.1)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | 1.6 (5.9) | -0.6 (8.4) | -0.6 (5.2) | 2.1 (6.5) | 6.7 (14.4)

21. Primary Outcome: Change From Study Baseline Over Time in Supine Systolic Blood Pressure
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
mmHg
  Study Baseline | 136.3 (12.9) | 136.3 (12.9) | 136.3 (12.9) | 133.9 (10.8) | 132.9 (10.9) | 132.9 (10.9)
  Change at Cycle Day 1, 0 h | -8.9 (9.9) | -9.8 (19.6) | -18.7 (16.4) | -16.1 (10.3) | -15.0 (14.3) | -16.1 (15.7)
  Change at Cycle Day 1, 1 h | -14.8 (13.0) | -18.1 (18.7) | -25.6 (16.8) | -24.0 (13.5) | -22.9 (13.2) | -27.2 (13.5)
  Change at Cycle Day 1, 2 h | -17.3 (11.5) | -22.5 (17.8) | -27.5 (15.7) | -27.9 (14.5) | -26.6 (16.8) | -27.2 (15.1)
  Change at Cycle Day 1, 4 h | -13.5 (10.7) | -18.4 (13.0) | -24.4 (13.4) | -23.9 (15.1) | -27.0 (14.7) | -25.3 (16.7)
  Change at Cycle Day 1, 8 h | -16.6 (12.0) | -17.7 (13.5) | -25.3 (11.5) | -21.7 (13.5) | -24.3 (14.4) | -30.6 (15.5)
  Change at Cycle Day 1, 12 h | -14.4 (12.7) | -15.5 (16.8) | -23.8 (13.4) | -20.9 (14.2) | -22.3 (15.6) | -23.4 (17.4)
  Change at Cycle Day 3, 0 h | -13.3 (15.0) | -13.0 (16.1) | -18.3 (16.1) | -18.5 (15.1) | -16.9 (11.5) | -18.8 (16.7)
  Change at Cycle Day 3, 1 h | -16.1 (15.6) | -22.1 (17.8) | -24.9 (21.1) | -26.3 (15.1) | -24.7 (16.3) | -25.7 (13.5)
  Change at Cycle Day 3, 2 h: number analyzed (Participants) | 10 | 11 | 11 | 10 | 9 | 9
  Change at Cycle Day 3, 2 h | -16.1 (15.5) | -23.2 (16.7) | -27.7 (18.7) | -28.8 (15.7) | -28.0 (12.8) | -26.6 (12.0)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | -15.4 (15.0) | -20.5 (14.6) | -23.5 (16.3) | -26.2 (12.5) | -24.9 (14.3) | -20.6 (13.5)

22. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in Supine Systolic Blood Pressure
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
mmHg
  Time Matched Baseline (Cycle Day 1, 0 h) | 127.4 (9.1) | 127.4 (9.1) | 126.3 (8.9) | 125.2 (8.7) | 125.2 (8.7)
  Change at Cycle Day 1, 0 h | -0.9 (14.0) | -9.8 (9.9) | -8.5 (7.9) | -7.3 (7.4) | -8.4 (11.8)
  Time Matched Baseline (Cycle Day 1, 1 h) | 121.5 (11.3) | 121.5 (11.3) | 121.2 (11.8) | 119.7 (11.5) | 119.7 (11.5)
  Change at Cycle Day 1, 1 h | -3.3 (12.1) | -10.8 (11.1) | -11.3 (10.6) | -9.7 (11.4) | -14.0 (11.5)
  Time Matched Baseline (Cycle Day 1, 2 h) | 119.0 (8.8) | 119.0 (8.8) | 117.6 (7.9) | 117.2 (8.3) | 117.2 (8.3)
  Change at Cycle Day 1, 2 h | -5.3 (11.4) | -10.3 (11.4) | -11.6 (7.5) | -10.9 (8.1) | -11.6 (6.8)
  Time Matched Baseline (Cycle Day 1, 4 h) | 122.7 (6.4) | 122.7 (6.4) | 121.8 (5.9) | 120.7 (4.9) | 120.7 (4.9)
  Change at Cycle Day 1, 4 h | -4.8 (8.8) | -10.8 (11.3) | -11.8 (11.6) | -14.8 (10.4) | -13.1 (10.4)
  Time Matched Baseline (Cycle Day 1, 8 h) | 119.6 (9.9) | 119.6 (9.9) | 117.3 (6.5) | 116.4 (6.3) | 116.4 (6.3)
  Change at Cycle Day 1, 8 h | -1.1 (12.8) | -8.6 (11.1) | -5.1 (11.4) | -7.9 (11.4) | -14.1 (9.3)
  Time Matched Baseline (Cycle Day 1, 12 h) | 121.9 (10.7) | 121.9 (10.7) | 120.7 (10.4) | 119.0 (9.5) | 119.0 (9.5)
  Change at Cycle Day 1, 12 h | -1.2 (13.7) | -9.5 (9.8) | -7.7 (10.7) | -8.4 (9.2) | -9.6 (12.5)
  Time Matched Baseline (Cycle Day 3, 0 h) | 123.0 (11.4) | 123.0 (11.4) | 124.0 (11.5) | 124.3 (12.1) | 124.3 (12.1)
  Change at Cycle Day 3, 0 h | 0.3 (11.3) | -5.0 (12.2) | -8.6 (10.8) | -8.3 (10.2) | -10.2 (16.6)
  Time Matched Baseline (Cycle Day 3, 1 h) | 120.2 (12.6) | 120.2 (12.6) | 121.0 (12.9) | 121.3 (13.7) | 121.3 (13.7)
  Change at Cycle Day 3, 1 h | -6.0 (7.9) | -8.8 (10.4) | -13.4 (11.3) | -13.1 (15.7) | -14.1 (10.6)
  Time Matched Baseline (Cycle Day 3, 2 h): number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Time Matched Baseline (Cycle Day 3, 2 h) | 119.2 (10.8) | 119.2 (10.8) | 119.4 (11.5) | 120.4 (11.9) | 120.4 (11.9)
  Change at Cycle Day 3, 2 h: number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Change at Cycle Day 3, 2 h | -5.5 (6.8) | -10.4 (6.0) | -13.9 (5.0) | -16.3 (9.5) | -14.8 (4.7)
  Time Matched Baseline (Cycle Day 3, 8 h): number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Time Matched Baseline (Cycle Day 3, 8 h) | 120.9 (12.0) | 120.9 (12.0) | 120.6 (13.2) | 122.1 (13.1) | 122.1 (13.1)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | -5.1 (10.3) | -8.1 (9.2) | -12.1 (10.6) | -14.1 (10.4) | -9.8 (13.9)

23. Primary Outcome: Change From Study Baseline Over Time in Supine Diastolic Blood Pressure
Description: Study baseline is defined as the Day -1 assessment.
Time Frame: as for outcome 19
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
mmHg
  Study Baseline | 80.4 (5.9) | 80.4 (5.9) | 80.4 (5.9) | 79.9 (6.0) | 78.2 (2.9) | 78.2 (2.9)
  Change at Cycle Day 1, 0 h | -3.3 (5.1) | -4.4 (9.2) | -6.9 (6.9) | -6.4 (6.8) | -6.3 (5.6) | -5.9 (6.1)
  Change at Cycle Day 1, 1 h | -6.8 (6.8) | -7.9 (8.4) | -12.5 (8.2) | -13.3 (7.0) | -11.3 (5.5) | -13.7 (6.0)
  Change at Cycle Day 1, 2 h | -8.4 (7.4) | -10.9 (9.4) | -12.9 (7.5) | -16.3 (8.2) | -11.7 (6.6) | -13.3 (5.9)
  Change at Cycle Day 1, 4 h | -8.2 (4.9) | -8.2 (7.3) | -10.1 (5.8) | -11.7 (6.6) | -12.0 (4.9) | -10.8 (5.5)
  Change at Cycle Day 1, 8 h | -7.2 (7.5) | -6.7 (8.7) | -11.5 (6.3) | -10.1 (8.8) | -8.4 (7.7) | -13.3 (6.8)
  Change at Cycle Day 1, 12 h | -6.5 (6.6) | -8.6 (8.7) | -9.7 (10.6) | -10.3 (9.7) | -9.9 (6.8) | -11.0 (9.4)
  Change at Cycle Day 3, 0 h | -4.6 (6.7) | -2.6 (6.9) | -5.6 (7.1) | -7.0 (6.5) | -7.4 (5.4) | -5.3 (6.8)
  Change at Cycle Day 3, 1 h | -7.6 (7.9) | -10.9 (9.1) | -14.1 (9.6) | -13.6 (8.8) | -13.3 (6.3) | -13.2 (6.3)
  Change at Cycle Day 3, 2 h: number analyzed (Participants) | 10 | 11 | 11 | 10 | 9 | 9
  Change at Cycle Day 3, 2 h | -4.8 (8.6) | -10.5 (8.9) | -13.5 (8.4) | -12.3 (10.7) | -12.2 (5.6) | -16.3 (5.3)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | -7.5 (7.8) | -9.1 (8.5) | -11.2 (6.2) | -12.1 (8.3) | -10.9 (5.3) | -9.4 (5.6)

24. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in Supine Diastolic Blood Pressure
Description: as for outcome 20
Time Frame: as for outcome 20
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
mmHg
  Time Matched Baseline (Cycle Day 1, 0 h) | 77.1 (5.3) | 77.1 (5.3) | 77.0 (5.6) | 75.7 (3.8) | 75.7 (3.8)
  Change at Cycle Day 1, 0 h | -1.1 (6.2) | -3.6 (3.7) | -3.5 (4.4) | -3.8 (2.5) | -3.3 (4.9)
  Time Matched Baseline (Cycle Day 1, 1 h) | 73.5 (8.0) | 73.5 (8.0) | 74.1 (8.2) | 72.1 (5.6) | 72.1 (5.6)
  Change at Cycle Day 1, 1 h | -1.1 (6.5) | -5.6 (7.4) | -7.5 (7.3) | -5.2 (5.3) | -7.6 (5.8)
  Time Matched Baseline (Cycle Day 1, 2 h) | 72.0 (5.5) | 72.0 (5.5) | 71.9 (5.8) | 71.4 (5.9) | 71.4 (5.9)
  Change at Cycle Day 1, 2 h | -2.5 (6.0) | -4.5 (5.4) | -8.3 (4.7) | -4.9 (6.8) | -6.6 (5.7)
  Time Matched Baseline (Cycle Day 1, 4 h) | 72.2 (6.1) | 72.2 (6.1) | 72.5 (6.4) | 71.0 (4.5) | 71.0 (4.5)
  Change at Cycle Day 1, 4 h | 0 (7.0) | -1.9 (6.1) | -4.3 (6.6) | -4.8 (6.0) | -3.6 (3.3)
  Time Matched Baseline (Cycle Day 1, 8 h) | 73.2 (7.3) | 73.2 (7.3) | 71.9 (6.2) | 70.9 (5.7) | 70.9 (5.7)
  Change at Cycle Day 1, 8 h | 0.5 (9.9) | -4.3 (8.4) | -2.1 (7.9) | -1.1 (10.6) | -6.0 (6.2)
  Time Matched Baseline (Cycle Day 1, 12 h) | 73.8 (7.7) | 73.8 (7.7) | 72.9 (7.4) | 71.3 (5.9) | 71.3 (5.9)
  Change at Cycle Day 1, 12 h | -2.1 (7.2) | -3.2 (10.7) | -3.3 (6.8) | -3.0 (5.4) | -4.1 (5.6)
  Time Matched Baseline (Cycle Day 3, 0 h) | 75.7 (4.3) | 75.7 (4.3) | 76.1 (4.4) | 75.7 (4.4) | 75.7 (4.4)
  Change at Cycle Day 3, 0 h | 2.0 (4.4) | -1.0 (4.8) | -3.2 (4.6) | -4.9 (3.3) | -2.8 (6.3)
  Time Matched Baseline (Cycle Day 3, 1 h) | 72.7 (6.1) | 72.7 (6.1) | 72.9 (6.3) | 72.6 (6.6) | 72.6 (6.6)
  Change at Cycle Day 3, 1 h | -3.3 (4.6) | -6.5 (6.0) | -6.6 (5.9) | -7.7 (7.3) | -7.6 (5.5)
  Time Matched Baseline (Cycle Day 3, 2 h): number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Time Matched Baseline (Cycle Day 3, 2 h) | 75.6 (6.3) | 75.6 (6.3) | 75.3 (6.7) | 75.4 (7.1) | 75.4 (7.1)
  Change at Cycle Day 3, 2 h: number analyzed (Participants) | 10 | 10 | 9 | 8 | 8
  Change at Cycle Day 3, 2 h | -5.1 (4.0) | -8.0 (6.4) | -7.0 (6.2) | -8.5 (4.9) | -13.3 (5.1)
  Time Matched Baseline (Cycle Day 3, 8 h): number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Time Matched Baseline (Cycle Day 3, 8 h) | 72.8 (6.5) | 72.8 (6.5) | 73.0 (6.8) | 73.0 (6.8) | 73.0 (6.8)
  Change at Cycle Day 3, 8 h: number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 8 h | -1.5 (5.5) | -3.6 (4.0) | -4.8 (5.3) | -5.7 (3.9) | -4.2 (5.5)

25. Primary Outcome: Orthostatic Pulse Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: Cycle Day 1, Predose; Cycle Day 1, 1 h; Cycle Day 1, 2 h; Cycle Day 1, 4 h; Cycle Day 1, 8 h; Cycle Day 1, 12 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
bpm
  Cycle Day 1, Predose | 9.7 (3.8) | 11.6 (5.6) | 11.0 (4.1) | 11.9 (3.8) | 11.0 (3.9) | 10.4 (2.7)
  Cycle Day 1, 1 h | 9.7 (5.4) | 11.5 (7.1) | 12.6 (6.4) | 17.8 (6.1) | 17.8 (7.6) | 16.0 (7.4)
  Cycle Day 1, 2 h | 10.9 (4.1) | 10.6 (5.9) | 12.3 (8.4) | 14.6 (6.8) | 13.9 (5.9) | 15.6 (5.7)
  Cycle Day 1, 4 h | 9.5 (7.7) | 10.3 (9.5) | 11.0 (6.4) | 14.6 (5.3) | 12.3 (9.3) | 14.8 (8.0)
  Cycle Day 1, 8 h | 10.8 (7.8) | 10.3 (6.7) | 12.7 (6.5) | 13.0 (3.4) | 15.2 (4.4) | 11.0 (7.6)
  Cycle Day 1, 12 h | 10.7 (4.8) | 10.6 (5.1) | 9.9 (13.0) | 10.8 (7.5) | 13.0 (7.4) | 11.3 (6.8)

26. Primary Outcome: Orthostatic Systolic Blood Pressure Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: Cycle Day 1, Predose; Cycle Day 1, 1 h; Cycle Day 1, 2 h; Cycle Day 1, 4 h; Cycle Day 1, 8 h; Cycle Day 1, 12 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
mmHg
  Cycle Day 1, Predose | 4.4 (7.2) | 3.7 (6.5) | 5.9 (7.3) | 4.0 (13.0) | 3.4 (5.3) | 4.2 (9.1)
  Cycle Day 1, 1 h | 7.0 (5.6) | 9.1 (8.4) | 5.2 (3.5) | 5.8 (8.2) | 4.0 (6.8) | 6.2 (6.7)
  Cycle Day 1, 2 h | 8.5 (12.4) | 8.2 (4.6) | 6.2 (8.7) | 7.3 (8.4) | 3.3 (6.5) | 4.6 (8.3)
  Cycle Day 1, 4 h | 3.6 (9.2) | 3.2 (8.7) | 4.2 (5.8) | 4.3 (5.0) | 6.3 (9.2) | 6.7 (7.7)
  Cycle Day 1, 8 h | 8.4 (5.8) | 5.4 (5.8) | 8.1 (14.1) | 5.5 (7.8) | 5.6 (4.9) | 8.0 (4.5)
  Cycle Day 1, 12 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Cycle Day 1, 12 h | 9.7 (10.5) | 6.2 (5.3) | 6.0 (6.1) | 8.0 (6.7) | 2.1 (4.5) | 3.4 (7.9)

27. Primary Outcome: Orthostatic Diastolic Blood Pressure Over Time
Description: An orthostatic measurement is obtained by subtracting the supine measurement from the standing measurement.
Time Frame: Cycle Day 1, Predose; Cycle Day 1, 1 h; Cycle Day 1, 2 h; Cycle Day 1, 4 h; Cycle Day 1, 8 h; Cycle Day 1, 12 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
mmHg
  Cycle Day 1, Predose | 7.0 (2.4) | 9.3 (4.7) | 8.1 (7.7) | 5.7 (5.1) | 8.3 (2.7) | 7.4 (4.4)
  Cycle Day 1, 1 h | 6.9 (4.1) | 7.0 (3.9) | 6.5 (3.7) | 4.7 (4.4) | 5.7 (3.6) | 5.8 (3.8)
  Cycle Day 1, 2 h | 10.5 (6.5) | 8.3 (3.5) | 6.5 (5.6) | 7.6 (3.7) | 3.2 (7.2) | 4.2 (4.6)
  Cycle Day 1, 4 h | 9.1 (3.6) | 6.6 (7.8) | 4.9 (4.3) | 5.1 (3.1) | 6.2 (2.7) | 6.9 (5.5)
  Cycle Day 1, 8 h | 9.1 (7.1) | 6.0 (5.5) | 7.9 (5.2) | 5.5 (3.4) | 4.7 (7.6) | 7.0 (5.0)
  Cycle Day 1, 12 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Cycle Day 1, 12 h | 8.6 (7.7) | 7.9 (3.9) | 5.5 (6.2) | 9.3 (6.3) | 6.6 (2.5) | 6.2 (4.3)

28. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in Ambulatory Blood Pressure Monitoring (ABPM) 4-Hour Averages of Systolic Blood Pressure
Description: Four-hour average is the average of ABPM assessments over 4 hours intervals from the time of dosing. Time-matched baseline is the 4 hours average during the placebo cycle (Day 2).
  Baseline is designated per protocol as Day 2 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 2 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2: 0-4 hrs, 4-8 hrs, 8-12 hrs
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0-4 hrs: Time Matched Baseline | 125.67 (10.39) | 125.67 (10.39) | 125.67 (10.39) | 125.72 (11.02) | 125.72 (11.02)
  0-4 hrs: Cycle Day 2 Change | -5.18 (5.70) | -10.57 (8.67) | -8.98 (9.08) | -11.57 (11.00) | -13.15 (12.59)
  4-8 hrs: Time Matched Baseline | 124.28 (8.07) | 124.28 (8.07) | 124.28 (8.07) | 123.32 (7.94) | 123.32 (7.94)
  4-8 hrs: Cycle Day 2 Change | -5.56 (10.61) | -9.45 (9.68) | -9.03 (12.55) | -13.26 (11.78) | -14.18 (10.07)
  8-12 hrs: Time Matched Baseline | 128.95 (9.99) | 128.95 (9.99) | 128.95 (9.99) | 127.42 (9.26) | 127.42 (9.26)
  8-12 hrs: Cycle Day 2 Change | -2.65 (12.85) | -8.80 (14.91) | -6.81 (10.27) | -10.51 (12.34) | -11.93 (13.47)

29. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 30 Minute Averages of Systolic Blood Pressure
Description: Thirty-minute average is the average of ABPM assessments over 30 minutes intervals from the time of dosing. Time-matched baseline is the 30 minutes average during the placebo cycle (Day 2).
  Baseline is designated per protocol as Day 2 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 2 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2: 0.5 hr, 1 hr, 1.5 hrs, 2 hrs, 2.5 hrs, 3 hrs, 3.5 hrs, 4 hrs, 4.5 hrs, 5 hrs, 5.5 hrs, 6 hrs, 6.5 hrs, 7 hrs, 7.5 hrs, 8 hrs, 8.5 hrs, 9 hrs, 9.5 hrs, 10 hrs, 10.5 hrs, 11 hrs, 11.5 hrs, 12 hrs
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0.5 hr: Time Matched Baseline | 140.30 (18.66) | 140.30 (18.66) | 140.30 (18.66) | 138.22 (18.53) | 138.22 (18.53)
  0.5 hr: Cycle Day 2 Change | -4.90 (6.89) | -14.80 (8.78) | -10.10 (10.09) | -11.67 (13.06) | -10.67 (9.95)
  1 hr: Time Matched Baseline | 128.60 (12.56) | 128.60 (12.56) | 128.60 (12.56) | 128.89 (13.29) | 128.89 (13.29)
  1 hr: Cycle Day 2 Change | -7.70 (12.36) | -12.50 (14.00) | -10.80 (16.19) | -8.56 (17.41) | -14.22 (15.74)
  1.5 hrs: Time Matched Baseline | 125.10 (13.99) | 125.10 (13.99) | 125.10 (13.99) | 125.67 (14.71) | 125.67 (14.71)
  1.5 hrs: Cycle Day 2 Change | -5.00 (11.75) | -9.10 (18.46) | -10.40 (14.39) | -14.33 (12.71) | -13.67 (16.81)
  2 hrs: Time Matched Baseline | 122.70 (10.68) | 122.70 (10.68) | 122.70 (10.68) | 123.22 (11.19) | 123.22 (11.19)
  2 hrs: Cycle Day 2 Change | -5.10 (14.42) | -6.30 (10.56) | -8.90 (9.92) | -12.56 (13.25) | -13.11 (16.32)
  2.5 hrs: Time Matched Baseline | 120.20 (6.05) | 120.20 (6.05) | 120.20 (6.05) | 120.22 (6.42) | 120.22 (6.42)
  2.5 hrs: Cycle Day 2 Change | 0 (13.55) | -10.10 (12.56) | -7.40 (12.81) | -13.11 (13.16) | -12.33 (12.11)
  3 hrs: Time Matched Baseline | 119.10 (13.04) | 119.10 (13.04) | 119.10 (13.04) | 118.78 (13.79) | 118.78 (13.79)
  3 hrs: Cycle Day 2 Change | -3.20 (16.29) | -6.40 (19.78) | -4.70 (17.61) | -8.22 (18.77) | -11.56 (18.42)
  3.5 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Time Matched Baseline | 120.89 (13.77) | 120.89 (13.77) | 120.89 (13.77) | 120.75 (14.71) | 120.75 (14.71)
  3.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Cycle Day 2 Change | -6.56 (15.95) | -14.11 (14.29) | -10.67 (12.36) | -9.25 (19.03) | -12.88 (22.40)
  4 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Time Matched Baseline | 126.30 (12.57) | 126.30 (12.57) | 123.78 (10.31) | 127.56 (12.65) | 127.56 (12.65)
  4 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Cycle Day 2 Change | -8.00 (8.94) | -11.30 (12.70) | -5.56 (13.31) | -13.78 (12.66) | -15.33 (18.41)
  4.5 hrs: Time Matched Baseline | 129.80 (13.60) | 129.80 (13.60) | 129.80 (13.60) | 127.33 (11.82) | 127.33 (11.82)
  4.5 hrs: Cycle Day 2 Change | -10.70 (11.98) | -10.50 (14.69) | -14.70 (10.71) | -8.78 (11.20) | -13.44 (17.40)
  5 hrs: Time Matched Baseline | 120.80 (14.44) | 120.80 (14.44) | 120.80 (14.44) | 119.56 (14.73) | 119.56 (14.73)
  5 hrs: Cycle Day 2 Change | -1.90 (13.89) | -6.20 (14.54) | -5.20 (19.86) | -7.33 (17.33) | -11.67 (17.43)
  5.5 hrs: Time Matched Baseline | 123.50 (16.18) | 123.50 (16.18) | 123.50 (16.18) | 123.33 (17.15) | 123.33 (17.15)
  5.5 hrs: Cycle Day 2 Change | -3.10 (15.74) | -9.40 (14.95) | -9.20 (14.90) | -18.11 (19.66) | -17.44 (20.73)
  6 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Time Matched Baseline | 122.00 (11.27) | 124.89 (7.01) | 122.00 (11.27) | 120.78 (11.23) | 120.78 (11.23)
  6 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Cycle Day 2 Change | -6.90 (16.04) | -12.00 (11.86) | -7.80 (13.80) | -15.33 (17.73) | -16.11 (14.48)
  6.5 hrs: Time Matched Baseline | 121.40 (7.68) | 121.40 (7.68) | 121.40 (7.68) | 121.44 (8.14) | 121.44 (8.14)
  6.5 hrs: Cycle Day 2 Change | -2.00 (17.95) | -7.60 (15.90) | -4.60 (17.60) | -12.44 (18.41) | -14.44 (13.97)
  7 hrs: Time Matched Baseline | 125.50 (10.17) | 125.50 (10.17) | 125.50 (10.17) | 126.22 (10.51) | 126.22 (10.51)
  7 hrs: Cycle Day 2 Change | -5.50 (13.88) | -11.60 (15.28) | -10.70 (16.34) | -15.44 (13.46) | -13.78 (11.36)
  7.5 hrs: Time Matched Baseline | 126.30 (12.31) | 126.30 (12.31) | 126.30 (12.31) | 125.44 (12.74) | 125.44 (12.74)
  7.5 hrs: Cycle Day 2 Change | -8.00 (16.80) | -12.30 (17.75) | -12.30 (21.43) | -16.56 (22.57) | -14.33 (20.27)
  8 hrs: Time Matched Baseline | 124.90 (12.68) | 124.90 (12.68) | 124.90 (12.68) | 122.44 (10.63) | 122.44 (10.63)
  8 hrs: Cycle Day 2 Change | -6.40 (21.29) | -9.10 (13.54) | -7.70 (19.81) | -12.11 (22.83) | -12.22 (15.70)
  8.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Time Matched Baseline | 126.10 (12.13) | 126.10 (12.13) | 125.11 (12.43) | 123.89 (10.52) | 123.89 (10.52)
  8.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Cycle Day 2 Change | -5.00 (13.32) | -8.40 (17.58) | -1.33 (9.42) | -12.11 (16.97) | -12.11 (17.51)
  9 hrs: Time Matched Baseline | 127.20 (11.12) | 127.20 (11.12) | 127.20 (11.12) | 125.67 (10.62) | 125.67 (10.62)
  9 hrs: Cycle Day 2 Change | -2.60 (17.44) | -7.90 (21.66) | -7.20 (18.33) | -13.78 (19.77) | -15.44 (15.16)
  9.5 hrs: Time Matched Baseline | 128.30 (14.38) | 128.30 (14.38) | 128.30 (14.38) | 126.78 (14.38) | 126.78 (14.38)
  9.5 hrs: Cycle Day 2 Change | -1.90 (23.19) | -14.00 (22.14) | -4.70 (18.69) | -12.11 (22.79) | -11.56 (19.64)
  10 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Time Matched Baseline | 128.56 (14.78) | 128.56 (14.78) | 128.56 (14.78) | 126.50 (14.36) | 126.50 (14.36)
  10 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Cycle Day 2 Change | -2.78 (20.11) | -10.67 (19.54) | -5.44 (13.42) | -9.63 (22.49) | -4.25 (24.81)
  10.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Time Matched Baseline | 136.90 (19.17) | 137.89 (20.07) | 136.90 (19.17) | 133.33 (16.45) | 133.33 (16.45)
  10.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Cycle Day 2 Change | -5.20 (22.09) | -5.78 (18.03) | -8.10 (16.13) | -11.33 (11.96) | -11.78 (16.28)
  11 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Time Matched Baseline | 133.44 (14.97) | 133.70 (14.13) | 133.44 (14.97) | 133.11 (14.86) | 133.11 (14.86)
  11 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Cycle Day 2 Change | -3.00 (16.05) | -15.50 (11.64) | -12.56 (9.17) | -15.78 (16.54) | -19.00 (21.04)
  11.5 hrs: Time Matched Baseline | 126.30 (10.04) | 126.30 (10.04) | 126.30 (10.04) | 126.11 (10.64) | 126.11 (10.64)
  11.5 hrs: Cycle Day 2 Change | -3.20 (8.40) | -3.20 (12.93) | -8.70 (6.06) | -4.56 (8.26) | -12.22 (14.01)
  12 hrs: Time Matched Baseline | 124.05 (9.42) | 124.05 (9.42) | 124.05 (9.42) | 123.17 (9.55) | 123.17 (9.55)
  12 hrs: Cycle Day 2 Change | 3.45 (9.54) | -4.10 (13.33) | -2.55 (10.93) | -4.94 (7.27) | -6.72 (14.85)

30. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM Daytime (12-Hour) Averages of Systolic Blood Pressure
Description: Daytime average is the average of ABPM assessments over 12 hours from the time of dosing. Time-matched baseline is the daytime average during the placebo cycle (Day 2).
  Baseline is designated per protocol as Day 2 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 2 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  Time-Matched Baseline | 126.27 (8.62) | 126.27 (8.62) | 126.27 (8.62) | 125.45 (8.72) | 125.45 (8.72)
  Cycle Day 2 Change | -4.42 (8.59) | -9.55 (9.98) | -8.22 (9.74) | -11.74 (10.71) | -13.05 (10.66)

31. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 4-Hour Averages of Diastolic Blood Pressure
Description: as for outcome 28
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2: 0-4 hrs, 4-8 hrs, 8-12 hrs
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0-4 hrs: Time Matched Baseline | 75.59 (6.05) | 75.59 (6.05) | 75.59 (6.05) | 74.94 (6.04) | 74.94 (6.04)
  0-4 hrs: Cycle Day 2 Change | -2.96 (3.75) | -7.59 (6.04) | -5.96 (5.53) | -7.94 (4.75) | -8.32 (6.28)
  4-8 hrs: Time Matched Baseline | 74.54 (7.54) | 74.54 (7.54) | 74.54 (7.54) | 72.88 (5.74) | 72.88 (5.74)
  4-8 hrs: Cycle Day 2 Change | -2.28 (7.46) | -4.03 (6.37) | -3.49 (8.91) | -7.61 (5.88) | -5.92 (7.12)
  8-12 hrs: Time Matched Baseline | 77.05 (6.31) | 77.05 (6.31) | 77.05 (6.31) | 75.75 (5.08) | 75.75 (5.08)
  8-12 hrs: Cycle Day 2 Change | 1.41 (5.71) | -3.70 (5.89) | -1.45 (4.79) | -4.63 (4.92) | -4.84 (6.78)

32. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 30 Minute Averages of Diastolic Blood Pressure
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0.5 hr: Time Matched Baseline | 87.90 (7.45) | 87.90 (7.45) | 87.90 (7.45) | 86.44 (6.21) | 86.44 (6.21)
  0.5 hr: Cycle Day 2 Change | -2.40 (6.04) | -8.70 (11.37) | -2.60 (6.50) | -7.56 (6.48) | -7.44 (9.81)
  1 hr: Time Matched Baseline | 77.90 (8.58) | 77.90 (8.58) | 77.90 (8.58) | 77.11 (8.71) | 77.11 (8.71)
  1 hr: Cycle Day 2 Change | -2.70 (7.29) | -10.40 (5.38) | -6.30 (10.63) | -7.56 (6.11) | -11.33 (8.08)
  1.5 hrs: Time Matched Baselline | 73.70 (11.02) | 73.70 (11.02) | 73.70 (11.02) | 72.89 (11.36) | 72.89 (11.36)
  1.5 hrs: Cycle Day 2 Change | -4.70 (11.54) | -6.30 (17.63) | -9.20 (10.61) | -9.78 (12.36) | -10.11 (10.76)
  2 hrs: Time Matched Baseline | 72.30 (7.59) | 72.30 (7.59) | 72.30 (7.59) | 71.00 (6.76) | 71.00 (6.76)
  2 hrs: Cycle Day 2 Change | -3.10 (8.54) | -5.60 (10.41) | -7.40 (8.37) | -5.33 (10.99) | -7.89 (9.40)
  2.5 hrs: Time Matched Baseline | 72.20 (7.93) | 72.20 (7.93) | 72.20 (7.93) | 71.89 (8.34) | 71.89 (8.34)
  2.5 hrs: Cycle Day 2 Change | -3.10 (12.91) | -9.70 (14.30) | -5.80 (11.59) | -11.11 (8.91) | -6.22 (9.90)
  3 hrs: Time Matched Baseline | 73.50 (11.83) | 73.50 (11.83) | 73.50 (11.83) | 73.44 (12.55) | 73.44 (12.55)
  3 hrs: Cycle Day 2 Change | -5.00 (9.82) | -7.90 (15.67) | -8.50 (14.18) | -8.44 (9.62) | -7.78 (17.50)
  3.5 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Time Matched Baseline | 70.33 (9.70) | 70.33 (9.70) | 70.33 (9.70) | 69.50 (10.01) | 69.50 (10.01)
  3.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Cycle Day 2 Change | -1.67 (12.57) | -6.89 (11.04) | -3.78 (9.19) | -8.00 (11.83) | -5.88 (13.89)
  4 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Time Matched Baseline | 76.60 (6.02) | 76.60 (6.02) | 76.33 (6.32) | 76.89 (6.31) | 76.89 (6.31)
  4 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Cycle Day 2 Change | -1.90 (6.40) | -6.10 (6.08) | -2.22 (11.02) | -6.56 (9.58) | -9.67 (9.71)
  4.5 hrs: Time Matched Baseline | 79.40 (12.88) | 79.40 (12.88) | 79.40 (12.88) | 76.56 (9.77) | 76.56 (9.77)
  4.5 hrs: Cycle Day 2 Change | -1.60 (11.72) | -5.80 (11.11) | -7.30 (9.78) | -3.78 (7.29) | -6.44 (7.84)
  5 hrs: Time Matched Baseline | 70.10 (14.10) | 70.10 (14.10) | 70.10 (14.10) | 67.78 (12.76) | 67.78 (12.76)
  5 hrs: Cycle Day 2 Change | -1.20 (14.65) | 1.70 (14.24) | -0.70 (13.49) | 0.11 (14.17) | -0.67 (14.49)
  5.5 hrs: Time Matched Baseline | 75.30 (7.54) | 75.30 (7.54) | 75.30 (7.54) | 74.22 (7.14) | 74.22 (7.14)
  5.5 hrs: Cycle Day 2 Change | -3.30 (9.19) | -6.00 (8.88) | -5.00 (7.62) | -14.67 (10.85) | -9.33 (9.63)
  6 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Time Matched Baseline | 74.80 (7.67) | 75.89 (7.27) | 74.80 (7.67) | 73.44 (6.75) | 73.44 (6.75)
  6 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Cycle Day 2 Change | -5.70 (16.38) | -7.44 (9.86) | -6.10 (10.87) | -15.22 (10.72) | -8.11 (10.45)
  6.5 hrs: Time Matched Baseline | 73.60 (7.17) | 73.60 (7.17) | 73.60 (7.17) | 72.67 (6.93) | 72.67 (6.93)
  6.5 hrs: Cycle Day 2 Change | -3.70 (12.28) | -5.30 (6.86) | -3.20 (14.86) | -8.00 (10.81) | -8.78 (12.34)
  7 hrs: Time Matched Baseline | 75.70 (7.76) | 75.70 (7.76) | 75.70 (7.76) | 74.67 (7.47) | 74.67 (7.47)
  7 hrs: Cycle Day 2 Change | -1.50 (10.56) | -5.60 (10.39) | -1.70 (12.46) | -11.22 (10.11) | -4.78 (11.98)
  7.5 hrs: Time Matched Baseline | 73.70 (12.29) | 73.70 (12.29) | 73.70 (12.29) | 71.89 (11.54) | 71.89 (11.54)
  7.5 hrs: Cycle Day 2 Change | -0.80 (12.65) | -3.50 (14.73) | -3.20 (16.51) | -2.78 (15.71) | -4.11 (20.57)
  8 hrs: Time Matched Baseline | 73.70 (13.28) | 73.70 (13.28) | 73.70 (13.28) | 71.78 (12.52) | 71.78 (12.52)
  8 hrs: Cycle Day 2 Change | -0.40 (15.46) | -1.80 (12.93) | -0.70 (13.56) | -5.33 (17.05) | -5.11 (18.45)
  8.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Time Matched Baseline | 73.70 (9.26) | 73.70 (9.26) | 73.33 (9.75) | 71.33 (5.79) | 71.33 (5.79)
  8.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Cycle Day 2 Change | 2.20 (9.85) | -3.60 (7.60) | 0.89 (10.48) | -2.67 (10.23) | -2.78 (11.22)
  9 hrs: Time Matched Baseline | 75.90 (10.34) | 75.90 (10.34) | 75.90 (10.34) | 74.22 (9.42) | 74.22 (9.42)
  9 hrs: Cycle Day 2 Change | 3.80 (11.51) | -0.90 (13.92) | -0.80 (12.86) | -6.67 (12.74) | -6.67 (12.13)
  9.5 hrs: Time Matched Baseline | 80.90 (10.28) | 80.90 (10.28) | 80.90 (10.28) | 80.00 (10.48) | 80.00 (10.48)
  9.5 hrs: Cycle Day 2 Change | 0.60 (13.48) | -12.20 (11.63) | -3.60 (15.04) | -9.78 (11.38) | -7.11 (13.36)
  10 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Time Matched Baseline | 79.56 (7.32) | 79.56 (7.32) | 79.56 (7.32) | 78.63 (7.23) | 78.63 (7.23)
  10 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Cycle Day 2 Change | 0.56 (10.45) | -3.67 (9.68) | -1.78 (4.66) | -7.75 (13.04) | -3.75 (12.69)
  10.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Time Matched Baseline | 83.60 (10.24) | 84.22 (10.66) | 83.60 (10.24) | 82.56 (10.28) | 82.56 (10.28)
  10.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Cycle Day 2 Change | -2.80 (9.38) | -4.56 (9.15) | -1.60 (4.88) | -8.11 (11.24) | -9.22 (10.10)
  11 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Time Matched Baseline | 76.22 (8.45) | 77.00 (8.34) | 76.22 (8.45) | 75.89 (8.02) | 75.89 (8.02)
  11 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Cycle Day 2 Change | 0.89 (10.56) | -5.40 (7.85) | -5.56 (8.00) | -6.44 (9.94) | -8.22 (12.08)
  11.5 hrs: Time Matched Baseline | 73.50 (9.96) | 73.50 (9.96) | 73.50 (9.96) | 72.78 (10.28) | 72.78 (10.28)
  11.5 hrs: Cycle Day 2 Change | 0.20 (9.50) | -0.50 (11.65) | -2.80 (8.07) | 0.78 (10.37) | -2.78 (10.29)
  12 hrs: Time Matched Baseline | 73.20 (6.44) | 73.20 (6.44) | 73.20 (6.44) | 71.56 (4.03) | 71.56 (4.03)
  12 hrs: Cycle Day 2 Change | 5.30 (8.21) | -0.10 (5.57) | 2.50 (12.06) | 1.89 (9.49) | 0.89 (8.37)

33. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM Daytime (12-Hour) Averages of Diastolic Blood Pressure
Description: Daytime average is the average of ABPM assessments over 12 hours from the time of dosing. Time-matched baseline is the daytime average during the placebo cycle (Day 2).
  Baseline is designated per protocol as Day 2 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment). To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 2 of each IW-1973 dose are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  Time-Matched Baseline | 75.71 (6.27) | 75.71 (6.27) | 75.71 (6.27) | 74.51 (5.28) | 74.51 (5.28)
  Cycle Day 2 Change | -1.26 (4.08) | -5.10 (4.67) | -3.59 (5.72) | -6.71 (4.38) | -6.34 (5.84)

34. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 4-Hour Averages of Mean Arterial Pressure
Description: as for outcome 28
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2: 0-4 hrs, 4-8 hrs, 8-12 hrs
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0-4 hrs: Time Matched Baseline | 92.61 (6.23) | 92.61 (6.23) | 92.61 (6.23) | 92.21 (6.47) | 92.21 (6.47)
  0-4 hrs: Cycle Day 2 Change | -3.93 (3.38) | -8.93 (6.29) | -7.64 (6.16) | -9.13 (6.21) | -9.67 (8.37)
  4-8 hrs: Time Matched Baseline | 91.38 (6.49) | 91.38 (6.49) | 91.38 (6.49) | 89.99 (5.06) | 89.99 (5.06)
  4-8 hrs: Cycle Day 2 Change | -3.50 (7.59) | -5.80 (6.58) | -5.55 (9.34) | -10.29 (6.73) | -8.65 (6.93)
  8-12 hrs: Time Matched Baseline | 93.99 (6.38) | 93.99 (6.38) | 93.99 (6.38) | 92.51 (4.63) | 92.51 (4.63)
  8-12 hrs: Cycle Day 2 Change | 0.36 (8.87) | -4.34 (7.72) | -3.00 (6.44) | -6.81 (5.80) | -6.58 (8.05)

35. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 30 Minute Averages of Mean Arterial Pressure
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0.5 hr: Time Matched Baseline | 104.50 (9.96) | 104.50 (9.96) | 104.50 (9.96) | 102.00 (6.42) | 102.00 (6.42)
  0.5 hr: Cycle Day 2 Change | -3.70 (7.21) | -9.20 (10.99) | -3.90 (8.50) | -5.33 (6.06) | -4.11 (10.41)
  1 hr: Time Matched Baseline | 96.80 (7.73) | 96.80 (7.73) | 96.80 (7.73) | 96.33 (8.05) | 96.33 (8.05)
  1 hr: Cycle Day 2 Change | -7.00 (7.73) | -12.70 (6.80) | -10.60 (11.05) | -10.11 (9.24) | -14.89 (9.31)
  1.5 hrs: Time Matched Baseline | 91.30 (13.02) | 91.30 (13.02) | 91.30 (13.02) | 91.22 (13.81) | 91.22 (13.81)
  1.5 hrs: Cycle Day 2 Change | -5.20 (11.39) | -8.80 (17.82) | -10.00 (11.55) | -11.67 (14.97) | -12.00 (15.28)
  2 hrs: Time Matched Baseline | 89.20 (6.58) | 89.20 (6.58) | 89.20 (6.58) | 88.44 (6.50) | 88.44 (6.50)
  2 hrs: Cycle Day 2 Change | -1.70 (11.16) | -6.10 (8.92) | -9.10 (8.52) | -8.11 (10.17) | -8.67 (16.51)
  2.5 hrs: Time Matched Baseline | 88.80 (6.70) | 88.80 (6.70) | 88.80 (6.70) | 88.67 (7.09) | 88.67 (7.09)
  2.5 hrs: Cycle Day 2 Change | -2.40 (12.75) | -11.40 (15.25) | -7.20 (10.94) | -12.22 (9.86) | -10.11 (9.83)
  3 hrs: Time Matched Baseline | 88.10 (11.24) | 88.10 (11.24) | 88.10 (11.24) | 88.22 (11.91) | 88.22 (11.91)
  3 hrs: Cycle Day 2 Change | -4.20 (10.54) | -6.90 (14.26) | -5.50 (15.17) | -8.78 (9.43) | -7.44 (17.26)
  3.5 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Time Matched Baseline | 87.44 (10.08) | 87.44 (10.08) | 87.44 (10.08) | 87.25 (10.75) | 87.25 (10.75)
  3.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Cycle Day 2 Change | -3.89 (13.40) | -9.00 (11.24) | -6.56 (8.80) | -8.63 (13.16) | -7.50 (15.68)
  4 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Time Matched Baseline | 94.10 (7.34) | 94.10 (7.34) | 92.78 (6.40) | 94.78 (7.45) | 94.78 (7.45)
  4 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Cycle Day 2 Change | -4.00 (8.46) | -7.90 (7.29) | -5.78 (10.33) | -8.78 (9.02) | -12.11 (13.60)
  4.5 hrs: Time Matched Baseline | 97.30 (10.92) | 97.30 (10.92) | 97.30 (10.92) | 94.67 (7.50) | 94.67 (7.50)
  4.5 hrs: Cycle Day 2 Change | -4.30 (7.75) | -7.40 (10.16) | -11.30 (8.14) | -5.89 (2.93) | -9.67 (7.94)
  5 hrs: Time Matched Baseline | 86.60 (12.47) | 86.60 (12.47) | 86.60 (12.47) | 84.56 (11.30) | 84.56 (11.30)
  5 hrs: Cycle Day 2 Change | -1.30 (14.03) | -0.80 (11.52) | -2.80 (15.51) | -3.00 (12.61) | -5.11 (12.29)
  5.5 hrs: Time Matched Baseline | 92.00 (7.21) | 92.00 (7.21) | 92.00 (7.21) | 91.11 (7.04) | 91.11 (7.04)
  5.5 hrs: Cycle Day 2 Change | -3.40 (10.95) | -8.70 (8.38) | -7.10 (8.12) | -18.44 (10.03) | -13.33 (11.09)
  6 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Time Matched Baseline | 90.70 (7.18) | 92.33 (5.29) | 90.70 (7.18) | 89.78 (6.96) | 89.78 (6.96)
  6 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Cycle Day 2 Change | -5.80 (14.99) | -9.00 (9.54) | -7.20 (11.06) | -15.56 (10.50) | -10.67 (11.15)
  6.5 hrs: Time Matched Baseline | 89.80 (6.41) | 89.80 (6.41) | 89.80 (6.41) | 89.44 (6.69) | 89.44 (6.69)
  6.5 hrs: Cycle Day 2 Change | -3.50 (12.09) | -6.10 (9.18) | -4.40 (12.82) | -11.44 (11.07) | -11.33 (10.63)
  7 hrs: Time Matched Baseline | 92.90 (7.92) | 92.90 (7.92) | 92.90 (7.92) | 92.44 (8.26) | 92.44 (8.26)
  7 hrs: Cycle Day 2 Change | -3.90 (12.06) | -8.50 (12.43) | -5.60 (12.73) | -14.11 (10.81) | -6.44 (11.67)
  7.5 hrs: Time Matched Baseline | 90.50 (11.72) | 90.50 (11.72) | 90.50 (11.72) | 88.78 (11.01) | 88.78 (11.01)
  7.5 hrs: Cycle Day 2 Change | -2.70 (15.60) | -3.90 (15.15) | -3.70 (17.84) | -6.33 (16.67) | -5.44 (18.26)
  8 hrs: Time Matched Baseline | 91.20 (13.00) | 91.20 (13.00) | 91.20 (13.00) | 89.11 (11.88) | 89.11 (11.88)
  8 hrs: Cycle Day 2 Change | -3.10 (17.12) | -3.90 (12.57) | -2.30 (15.82) | -7.56 (17.98) | -7.22 (13.63)
  8.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Time Matched Baseline | 91.80 (10.08) | 91.80 (10.08) | 91.00 (10.34) | 89.44 (7.20) | 89.44 (7.20)
  8.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Cycle Day 2 Change | -0.80 (11.21) | -6.30 (9.26) | -0.89 (10.29) | -6.11 (12.73) | -6.33 (11.28)
  9 hrs: Time Matched Baseline | 92.00 (8.50) | 92.00 (8.50) | 92.00 (8.50) | 90.44 (7.35) | 90.44 (7.35)
  9 hrs: Cycle Day 2 Change | 3.30 (12.00) | -1.80 (14.61) | -1.30 (14.25) | -7.44 (12.41) | -8.11 (11.26)
  9.5 hrs: Time Matched Baseline | 96.40 (11.75) | 96.40 (11.75) | 96.40 (11.75) | 95.22 (11.82) | 95.22 (11.82)
  9.5 hrs: Cycle Day 2 Change | 1.50 (20.74) | -11.90 (14.81) | -3.40 (16.81) | -11.11 (15.32) | -8.22 (16.05)
  10 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Time Matched Baseline | 95.11 (9.68) | 95.11 (9.68) | 95.11 (9.68) | 93.63 (9.18) | 93.63 (9.18)
  10 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Cycle Day 2 Change | -0.44 (14.79) | -4.89 (10.73) | -2.56 (7.99) | -9.75 (14.32) | -2.50 (18.24)
  10.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Time Matched Baseline | 101.00 (10.84) | 101.78 (11.20) | 101.00 (10.84) | 98.89 (9.06) | 98.89 (9.06)
  10.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Cycle Day 2 Change | -2.70 (13.15) | -3.67 (10.95) | -3.50 (6.52) | -10.11 (7.69) | -10.67 (11.45)
  11 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Time Matched Baseline | 95.00 (10.28) | 95.50 (9.82) | 95.00 (10.28) | 94.33 (9.66) | 94.33 (9.66)
  11 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Cycle Day 2 Change | -0.56 (11.17) | -7.10 (11.26) | -8.22 (9.92) | -10.00 (14.24) | -11.78 (14.70)
  11.5 hrs: Time Matched Baseline | 90.10 (8.45) | 90.10 (8.45) | 90.10 (8.45) | 89.56 (8.78) | 89.56 (8.78)
  11.5 hrs: Cycle Day 2 Change | -1.40 (7.66) | 0.60 (10.62) | -5.20 (5.39) | -0.78 (8.35) | -3.89 (7.46)
  12 hrs: Time Matched Baseline | 90.45 (6.30) | 90.45 (6.30) | 90.45 (6.30) | 88.94 (4.37) | 88.94 (4.37)
  12 hrs: Cycle Day 2 Change | 3.80 (7.63) | -0.25 (7.67) | 0.95 (10.96) | -0.72 (6.64) | -0.89 (7.88)

36. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM Daytime (12-Hour) Averages of Mean Arterial Pressure
Description: as for outcome 33
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  Time-Matched Baseline | 92.64 (5.77) | 92.64 (5.77) | 92.64 (5.77) | 91.55 (4.90) | 91.55 (4.90)
  Cycle Day 2 Change | -2.33 (5.21) | -6.33 (5.44) | -5.34 (6.58) | -8.72 (5.43) | -8.28 (6.54)

37. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 4-Hour Averages of Pulse
Description: as for outcome 28
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2: 0-4 hrs, 4-8 hrs, 8-12 hrs
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0-4 hrs: Time Matched Baseline | 75.61 (12.37) | 75.61 (12.37) | 75.61 (12.37) | 76.59 (12.70) | 76.59 (12.70)
  0-4 hrs: Cycle Day 2 Change | 2.49 (3.62) | 6.11 (4.49) | 8.91 (7.60) | 7.10 (4.43) | 7.38 (6.58)
  4-8 hrs: Time Matched Baseline | 73.24 (11.19) | 73.24 (11.19) | 73.24 (11.19) | 73.81 (11.72) | 73.81 (11.72)
  4-8 hrs: Cycle Day 2 Change | 9.24 (5.30) | 7.56 (6.51) | 6.50 (7.82) | 12.82 (7.16) | 8.89 (8.83)
  8-12 hrs: Time Matched Baseline | 76.22 (12.59) | 76.22 (12.59) | 76.22 (12.59) | 76.95 (13.13) | 76.95 (13.13)
  8-12 hrs: Cycle Day 2 Change | 1.91 (7.04) | -1.20 (6.52) | 1.51 (5.34) | 2.53 (5.55) | 3.35 (8.48)

38. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM 30 Minute Averages of Pulse
Description: as for outcome 29
Time Frame: as for outcome 29
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  0.5 hr: Time Matched Baseline | 76.30 (9.89) | 76.30 (9.89) | 76.30 (9.89) | 75.67 (10.27) | 75.67 (10.27)
  0.5 hr: Cycle Day 2 Change | -0.60 (4.17) | 1.60 (5.23) | 1.50 (8.34) | 2.67 (9.62) | 2.11 (5.42)
  1 hr: Time Matched Baseline | 73.50 (11.69) | 73.50 (11.69) | 73.50 (11.69) | 74.44 (11.99) | 74.44 (11.99)
  1 hr: Cycle Day 2 Change | 3.00 (6.09) | 7.30 (8.19) | 11.00 (10.09) | 8.11 (7.85) | 9.89 (9.98)
  1.5 hrs: Time Matched Baseline | 74.80 (12.25) | 74.80 (12.25) | 74.80 (12.25) | 75.56 (12.74) | 75.56 (12.74)
  1.5 hrs: Cycle Day 2 Change | 5.60 (4.93) | 18.90 (12.72) | 14.60 (14.21) | 10.44 (7.75) | 14.44 (5.39)
  2 hrs: Time Matched Baseline | 78.80 (15.30) | 78.80 (15.30) | 78.80 (15.30) | 80.22 (15.51) | 80.22 (15.51)
  2 hrs: Cycle Day 2 Change | 0.90 (8.13) | 7.40 (5.91) | 6.90 (7.03) | 14.00 (22.92) | 5.33 (9.50)
  2.5 hrs: Time Matched Baseline | 76.60 (13.43) | 76.60 (13.43) | 76.60 (13.43) | 77.89 (13.57) | 77.89 (13.57)
  2.5 hrs: Cycle Day 2 Change | 3.20 (7.79) | 5.20 (6.71) | 9.30 (12.28) | 8.44 (7.70) | 6.67 (11.70)
  3 hrs: Time Matched Baseline | 77.10 (15.53) | 77.10 (15.53) | 77.10 (15.53) | 78.56 (15.73) | 78.56 (15.73)
  3 hrs: Cycle Day 2 Change | 2.70 (9.01) | 1.20 (10.81) | 12.10 (14.56) | 2.22 (8.77) | 7.89 (12.23)
  3.5 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Time Matched Baseline | 74.33 (15.84) | 74.33 (15.84) | 74.33 (15.84) | 75.75 (16.31) | 75.75 (16.31)
  3.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  3.5 hrs: Cycle Day 2 Change | 2.78 (6.85) | 2.44 (5.17) | 8.33 (10.10) | 5.13 (10.52) | 5.13 (13.82)
  4 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Time Matched Baseline | 73.70 (15.98) | 73.70 (15.98) | 74.67 (16.64) | 75.11 (16.27) | 75.11 (16.27)
  4 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  4 hrs: Cycle Day 2 Change | 2.70 (6.63) | 3.90 (9.45) | 8.89 (13.59) | 5.78 (8.76) | 7.44 (13.53)
  4.5 hrs: Time Matched Baseline | 80.80 (13.73) | 80.80 (13.73) | 80.80 (13.73) | 81.56 (14.34) | 81.56 (14.34)
  4.5 hrs: Cycle Day 2 Change | 4.70 (7.02) | 2.70 (8.03) | 9.60 (15.24) | 10.56 (10.86) | 7.33 (9.64)
  5 hrs: Time Matched Baseline | 75.50 (10.21) | 75.50 (10.21) | 75.50 (10.21) | 76.44 (10.36) | 76.44 (10.36)
  5 hrs: Cycle Day 2 Change | 5.50 (11.45) | 7.90 (13.87) | 4.00 (10.65) | 17.78 (14.81) | 7.00 (15.26)
  5.5 hrs: Time Matched Baseline | 75.50 (10.10) | 75.50 (10.10) | 75.50 (10.10) | 76.11 (10.52) | 76.11 (10.52)
  5.5 hrs: Cycle Day 2 Change | 7.80 (11.69) | 5.70 (11.79) | 6.80 (11.12) | 10.00 (11.22) | 5.00 (13.22)
  6 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Time Matched Baseline | 72.00 (11.11) | 71.44 (11.63) | 72.00 (11.11) | 72.22 (11.76) | 72.22 (11.76)
  6 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  6 hrs: Cycle Day 2 Change | 12.60 (15.07) | 7.89 (9.57) | 7.40 (10.36) | 16.00 (13.87) | 8.56 (8.79)
  6.5 hrs: Time Matched Baseline | 71.40 (11.04) | 71.40 (11.04) | 71.40 (11.04) | 71.56 (11.70) | 71.56 (11.70)
  6.5 hrs: Cycle Day 2 Change | 13.10 (7.53) | 10.30 (10.47) | 8.30 (11.73) | 13.44 (10.57) | 13.00 (15.73)
  7 hrs: Time Matched Baseline | 69.10 (13.47) | 69.10 (13.47) | 69.10 (13.47) | 69.56 (14.20) | 69.56 (14.20)
  7 hrs: Cycle Day 2 Change | 14.00 (6.39) | 14.20 (14.20) | 8.30 (7.04) | 12.56 (4.42) | 13.00 (9.75)
  7.5 hrs: Time Matched Baseline | 70.40 (14.42) | 70.40 (14.42) | 70.40 (14.42) | 70.56 (15.28) | 70.56 (15.28)
  7.5 hrs: Cycle Day 2 Change | 9.70 (9.23) | 6.40 (8.76) | 5.70 (7.24) | 12.78 (9.76) | 11.67 (14.98)
  8 hrs: Time Matched Baseline | 71.20 (13.72) | 71.20 (13.72) | 71.20 (13.72) | 72.44 (13.94) | 72.44 (13.94)
  8 hrs: Cycle Day 2 Change | 6.50 (7.04) | 3.70 (5.14) | 1.90 (6.57) | 9.44 (8.11) | 5.56 (8.71)
  8.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Time Matched Baseline | 70.40 (13.63) | 70.40 (13.63) | 71.33 (14.12) | 71.22 (14.19) | 71.22 (14.19)
  8.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 10 | 9 | 9 | 9
  8.5 hrs: Cycle Day 2 Change | 5.80 (9.61) | 3.60 (7.18) | 1.33 (8.44) | 6.33 (7.92) | 8.78 (10.35)
  9 hrs: Time Matched Baseline | 71.30 (15.10) | 71.30 (15.10) | 71.30 (15.10) | 71.89 (15.89) | 71.89 (15.89)
  9 hrs: Cycle Day 2 Change | 5.30 (12.45) | 1.50 (9.65) | 1.60 (10.27) | 2.22 (13.89) | 4.44 (11.26)
  9.5 hrs: Time Matched Baseline | 72.00 (14.83) | 72.00 (14.83) | 72.00 (14.83) | 72.67 (15.57) | 72.67 (15.57)
  9.5 hrs: Cycle Day 2 Change | 3.60 (9.38) | 0.80 (9.20) | 3.60 (12.33) | 6.22 (7.51) | 8.78 (10.17)
  10 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Time Matched Baseline | 73.56 (12.82) | 73.56 (12.82) | 73.56 (12.82) | 74.13 (13.58) | 74.13 (13.58)
  10 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 9 | 9 | 8 | 8
  10 hrs: Cycle Day 2 Change | 4.89 (12.20) | 1.56 (8.00) | 3.11 (5.88) | 7.88 (9.60) | 5.75 (12.13)
  10.5 hrs: Time Matched Baseline: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Time Matched Baseline | 81.00 (12.12) | 81.78 (12.59) | 81.00 (12.12) | 81.33 (12.81) | 81.33 (12.81)
  10.5 hrs: Cycle Day 2 Change: number analyzed (Participants) | 10 | 9 | 10 | 9 | 9
  10.5 hrs: Cycle Day 2 Change | 0.60 (10.84) | -3.89 (10.17) | -1.00 (5.77) | 3.11 (11.19) | 2.11 (9.51)
  11 hrs: Time Matched Baseline: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Time Matched Baseline | 82.22 (17.10) | 81.30 (16.38) | 82.22 (17.10) | 82.56 (16.86) | 82.56 (16.86)
  11 hrs: Cycle Day 2 Change: number analyzed (Participants) | 9 | 10 | 9 | 9 | 9
  11 hrs: Cycle Day 2 Change | -4.33 (14.96) | -7.30 (14.62) | -2.67 (12.47) | -2.22 (15.21) | -3.56 (7.49)
  11.5 hrs: Time Matched Baseline | 81.60 (15.90) | 81.60 (15.90) | 81.60 (15.90) | 82.78 (16.40) | 82.78 (16.40)
  11.5 hrs: Cycle Day 2 Change | -3.10 (8.70) | -5.80 (11.28) | 0.20 (9.44) | -4.89 (9.52) | -3.56 (13.42)
  12 hrs: Time Matched Baseline | 78.45 (12.16) | 78.45 (12.16) | 78.45 (12.16) | 78.94 (12.79) | 78.94 (12.79)
  12 hrs: Cycle Day 2 Change | 2.25 (12.76) | 0.65 (9.60) | 4.40 (7.17) | 2.44 (6.94) | 2.78 (10.60)

39. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in ABPM Daytime (12-Hour) Averages of Pulse
Description: as for outcome 33
Time Frame: Time-Matched Baseline (Placebo Cycle); Cycle Day 2
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 10 | 10 | 10 | 9 | 9
mmHg
  Time-Matched Baseline | 75.01 (11.95) | 75.01 (11.95) | 75.01 (11.95) | 75.78 (12.42) | 75.78 (12.42)
  Cycle Day 2 Change | 4.55 (4.43) | 4.14 (4.80) | 5.70 (6.22) | 7.49 (3.88) | 6.55 (7.30)

40. Primary Outcome: Change From Pre- to Post-Nitroglycerin Dose Assessment in Supine Pulse
Time Frame: Follow-up Visit Day 32 (± 2 days)
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | All Participants
Number analyzed (Participants) | 11
bpm | -2.5 (5.4)

41. Primary Outcome: Change From Pre- to Post-Nitroglycerin Dose Assessment in Supine Systolic Blood Pressure
Time Frame: Follow-up Visit Day 32 (± 2 days)
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 11
mmHg | 3.5 (7.3)

42. Primary Outcome: Change From Pre- to Post-Nitroglycerin Dose Assessment in Supine Diastolic Blood Pressure
Time Frame: Follow-up Visit Day 32 (± 2 days)
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Participants
Number analyzed (Participants) | 11
mmHg | -0.5 (3.8)

43. Primary Outcome: Change From Study Baseline Over Time in Endothelial Function: Reactive Hyperemia Index (RHI)
Description: Study baseline is defined as the Day -1 assessment.
  Endothelial function was assessed by RHI value determined using the noninvasive EndoPAT™ (Itamar Medical; Caesarea, Israel) device. RHI is a validated measure of endothelial function, with a higher RHI indicating better endothelial function compared to a lower value. The full EndoPAT 2000 user manual (software version 3.7.x) recommends using RHI values >1.67 as a cutoff for normal endothelial function, with values ≤1.67 indicating endothelial dysfunction.
Time Frame: Study Baseline; Cycle Day 3: 0 h, 4 h, 12 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 11 | 10 | 9 | 9
units on a scale
  Study Baseline: number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 9
  Study Baseline | 2.21 (0.62) | 2.21 (0.62) | 2.28 (0.61) | 2.21 (0.66) | 2.28 (0.66) | 2.28 (0.66)
  Change at Cycle Day 3, 0 h: number analyzed (Participants) | 11 | 11 | 10 | 10 | 9 | 9
  Change at Cycle Day 3, 0 h | -0.08 (0.74) | -0.14 (0.91) | -0.13 (0.69) | 0.31 (1.08) | 0.20 (0.87) | -0.09 (0.87)
  Change at Cycle Day 3, 4 h | -0.39 (0.65) | 0.08 (0.99) | 0.01 (0.75) | -0.15 (0.80) | -0.17 (0.98) | -0.06 (0.78)
  Change at Cycle Day 3, 12 h: number analyzed (Participants) | 11 | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 12 h | -0.03 (0.64) | 0.33 (1.07) | 0.29 (0.68) | 0.07 (0.91) | 0.17 (1.06) | 0.37 (1.14)

44. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) Over Time in Endothelial Function: RHI
Description: Time-matched baseline for each timepoint is defined as the corresponding assessment during the placebo cycle.
  Endothelial function was assessed by RHI value determined using the noninvasive EndoPAT™ (Itamar Medical; Caesarea, Israel) device. RHI is a validated measure of endothelial function, with a higher RHI indicating better endothelial function compared to a lower value. The full EndoPAT 2000 user manual (software version 3.7.x) recommends using RHI values >1.67 as a cutoff for normal endothelial function, with values ≤1.67 indicating endothelial dysfunction.
  Baseline is designated per protocol as Day 3 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 3 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-matched Baseline (Placebo Cycle); Cycle Day 3: 0 h, 4 h, 12 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
units on a scale
  Time-Matched Baseline, 0 h: number analyzed (Participants) | 11 | 10 | 10 | 9 | 9
  Time-Matched Baseline, 0 h | 2.13 (0.57) | 2.15 (0.60) | 2.24 (0.49) | 2.28 (0.50) | 2.28 (0.50)
  Change at Cycle Day 3, 0 h: number analyzed (Participants) | 11 | 10 | 10 | 9 | 9
  Change at Cycle Day 3, 0 h | -0.07 (0.74) | 0 (0.87) | 0.28 (0.64) | 0.19 (0.39) | -0.09 (1.01)
  Time-Matched Baseline, 4 h | 1.82 (0.26) | 1.82 (0.26) | 1.82 (0.27) | 1.84 (0.27) | 1.84 (0.27)
  Change at Cycle Day 3, 4 h | 0.47 (1.02) | 0.40 (0.50) | 0.25 (0.60) | 0.26 (0.67) | 0.37 (0.75)
  Time-Matched Baseline, 12 h | 2.18 (0.48) | 2.18 (0.48) | 2.16 (0.51) | 2.12 (0.51) | 2.12 (0.51)
  Change at Cycle Day 3, 12 h: number analyzed (Participants) | 11 | 11 | 9 | 9 | 9
  Change at Cycle Day 3, 12 h | 0.36 (0.77) | 0.32 (0.39) | 0.20 (0.54) | 0.32 (0.66) | 0.53 (0.68)

45. Primary Outcome: Change From Pre- to Post-Nitroglycerin Dose Assessment in Endothelial Function: RHI
Description: Endothelial function was assessed by RHI value determined using the noninvasive EndoPAT™ (Itamar Medical; Caesarea, Israel) device. RHI is a validated measure of endothelial function, with a higher RHI indicating better endothelial function compared to a lower value. The full EndoPAT 2000 user manual (software version 3.7.x) recommends using RHI values >1.67 as a cutoff for normal endothelial function, with values ≤1.67 indicating endothelial dysfunction.
Time Frame: Follow-up Visit Day 32 (± 2 days)
Population: PD Population: all participants who received ≥1 dose of study drug and had ≥1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 11
units on a scale | -0.05 (0.37)

46. Primary Outcome: Change From Time-Matched Baseline (Placebo Cycle) in Platelet Function Assessments: Collagen/Epinephrine Time to Aggregation
Description: Time-matched baseline is defined as the corresponding assessment on Day 1 of the placebo cycle.
  Platelet function assessment used the PFA-100® instrument to evaluate collagen/epinephrine time to aggregation.
  Baseline is designated per protocol as Day 1 of the placebo cycle (Days 1-3; i.e., the first cycle of treatment) at given time point. To present 'change from time-matched baseline' endpoints, the values for time-matched baseline are presented as the first row of data, and the changes at Day 1 of each IW-1973 dose at given time point are presented as the second row of data.
Time Frame: Time-Matched Baseline (Placebo Cycle), Cycle Day 1, 0 h, Cycle Day 1, 4 h
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: secs
Arm/Group | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
Number analyzed (Participants) | 11 | 11 | 10 | 9 | 9
secs
  Time-Matched Baseline, 0 h: number analyzed (Participants) | 11 | 10 | 10 | 9 | 9
  Time-Matched Baseline, 0 h | 131.8 (60.6) | 132.8 (63.8) | 115.5 (28.7) | 114.8 (30.3) | 114.8 (30.3)
  Change at Cycle Day 1, 0 h: number analyzed (Participants) | 11 | 10 | 10 | 9 | 9
  Change at Cycle Day 1, 0 h | -21.0 (54.6) | -38.7 (46.5) | -6.8 (25.0) | 9.9 (47.4) | -4.2 (28.8)
  Time-Matched Baseline, 4 h | 121.3 (35.0) | 121.3 (35.0) | 115.0 (29.6) | 114.6 (31.4) | 114.6 (31.4)
  Change at Cycle Day 1, 4 h: number analyzed (Participants) | 11 | 11 | 10 | 9 | 8
  Change at Cycle Day 1, 4 h | -3.8 (22.2) | -15.5 (40.2) | -7.4 (23.9) | 14.2 (42.7) | -4.0 (32.4)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through end of trial (Day 46 [±3 days])
Description: Treatment emergent adverse events (TEAEs) are presented. TEAEs are defined as those AEs that started or worsened in severity after the initiation of study drug administration.
Arm/Group | Control | 10 mg IW-1973 | 20 mg IW-1973 | 30 mg IW-1973 | 40 mg IW-1973 | 50 mg IW-1973
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/10 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/10 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/11 | 3/11 | 2/11 | 4/10 | 3/9 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=11) | 10 mg IW-1973 (N=11) | 20 mg IW-1973 (N=11) | 30 mg IW-1973 (N=10) | 40 mg IW-1973 (N=9) | 50 mg IW-1973 (N=9)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tongue eruption (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure systolic decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
No separate placebo control. 2 of 11 enrolled participants discontinued prematurely. Participants were confined, diet and activity controlled. Multiple dose-escalation design had no washout period between dose cycles. EndoPAT device was exploratory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (2):
  • Study Protocol (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT02906579/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT02906579/SAP_001.pdf